CLINICAL TRIAL: NCT06274541
Title: Upfront Systematic Tumour BRCA Testing in Patients With High Grade Serous or Endometrioid Ovarian, Fallopian Tube or Primary Peritoneal Cancer: The t-BRCA Study
Brief Title: Upfront Systematic Tumour BRCA Testing in Patients With High Grade Serous or Endometrioid Ovarian, Fallopian Tube or Primary Peritoneal Cancer (HGSEC): The t-BRCA Study
Status: Active, not recruiting | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: CTRIAL-IE 18-01
Record Dates: First submitted 2019-06-06; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Serous Ovarian Tumor; Endometrioid Carcinoma Ovary; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Diploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HGSEC
  Interventions: Genetic: Somatic and Germline BRCA1/2 Testing

INTERVENTIONS:
Genetic: Somatic and Germline BRCA1/2 Testing — Germline BRCA1/2 mutation testing will be undertaken by NGS using blood samples. Somatic BRCA1/2 mutation testing will be undertaken by NGS using tumour tissue.

SUMMARY:
A pilot study to evaluate the feasibility of a NGS-based tumour BRCA1/2 mutation testing pathway initiated in the oncology clinic for patients with HGSEC, either at primary diagnosis or first relapse, whereby only patients with a positive germline BRCA1/2 mutation test will be referred to clinical genetics.

DETAILED DESCRIPTION:
This pilot study will evaluate the feasibility of a NGS-based tumour BRCA1/2 mutation testing pathway initiated in the oncology clinic for patients with HGSEC, either at primary diagnosis or first relapse, whereby only patients with a positive germline BRCA1/2 mutation test will be referred to clinical genetics. Germline BRCA1 and BRCA2 MLPA will be carried out to ensure accurate detection of BRCA1/2 LGRs. Patients with a high clinical risk of being germline mutation carriers and a negative germline BRCA1/2 mutation test should also be referred to clinical genetics. The investigators believe an upfront tumour testing pathway would be more cost-effective, as it would involve testing all patients for tumour BRCA1/2 mutations, followed by a single site germline test to clarify somatic/germline status of this mutation in approximately 25% of patients. In contrast, an upfront germline testing pathway would involve germline BRCA1/2 testing for all patients, followed by tumour BRCA1/2 tests in those 80 - 82% patients who do not have a germline BRCA1/2 mutation.

Systematic testing of patients in the oncology clinic for tumour BRCA1/2 mutations should not only ensure that all patients who are eligible for and agreeable to testing receive it, but also improve the quality of referrals to the clinical genetics team. Moreover, this approach is likely to significantly improve the identification rate of HGSEC patients with germline BRCA1/2 mutations, with resultant benefits for these patients in terms of cancer treatment and prevention, and their families in terms of opportunities for cancer prevention. The identification of patients with BRCA1/2 mutant HGSEC may facilitate treatment with effective maintenance therapies, or participation in clinical trials targeted at patients with BRCA1/2-mutated HGSEC. The incorporation of a health economics analysis relating to the introduction of this proposed testing pathway will further inform on the feasibility of its adoption into routine clinical practice on study completion. Finally, this study will also report on the currently unknown frequency, characteristics, disease course, and treatment patterns of germline and somatic BRCA1/2 mutations in an Irish population with HGSEC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high grade serous or high grade endometrioid ovarian, fallopian tube or primary peritoneal carcinoma who:

   Are newly diagnosed FIGO stage I - IV or Are currently undergoing primary chemotherapy +/- surgery or Are in remission after completing primary treatment for FIGO stage I - IV disease or Are being planned for, are undergoing or have completed treatment for first relapse
2. Patients with available tumour tissue (archival FFPE surgical resection or tissue/peritoneal biopsy) obtained prior to chemotherapy delivery, for tumour BRCA1/2 testing
3. Patients able to give signed and written informed consent
4. Patients aged 18 years and above

Exclusion Criteria:

1. Patients with non-high grade serous or non-high grade endometrioid ovarian, fallopian tube or primary peritoneal carcinoma or unclear histology
2. Patients in second or later relapse of their disease
3. Patients who are known BRCA1 or BRCA2 mutation carriers
4. Patients who have been previously tested for germline BRCA1/2 mutations or have been tested with a hereditary cancer gene panel.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with high grade serous or endometrioid ovarian, fallopian tube or primary peritoneal cancer (HGSEC), either at primary diagnosis or first relapse.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of an upfront BRCA1/2 mutation testing pathway in HGSEC in terms of clinicians' experience. | 24 months
  The primary outcome measure is to assess the feasibility and potential resource impact of the initiation of an ovarian cancer tumour tissue BRCA1/2 mutation testing pathway in the oncology clinic. This will be assessed in terms of clinicians' and patients' experience, impact on patient management and health economic analysis is the primary outcome measure. The primary outcome measure will be assessed via Clinician and patient questionnaires which will evaluate satisfaction/experience with tBRCA testing pathway.
Feasibility of an upfront BRCA1/2 mutation testing pathway in HGSEC in terms of patients' experience. | 24 months
  The feasibility will be assessed via Patient experience questionnaires. The patient experience questionnaires will evaluate patients' understanding of tBRCA testing, satisfaction/experience with tBRCA testing pathway, and feedback on the tBRCA testing pathway.
The impact on patient management by determining changes in patient treatment (use of a PARP inhibitor or enrolment in BRCA-targeted clinical trials). | 24 months
  A quantifiable outcome measure cannot be added here. The result of the BRCA testing impacts on the treatment decisions which the clinicians makes for the patient.
The impact on patient management by use of clinical genetics counselling sessions. | 24 months
The economic impact of implementing an upfront tumour BRCA1/2 mutation testing pathway in the oncology clinic for HGSEC on the Irish healthcare system, using a health economic analysis (decision analysis model) | 24 months
  A decision analysis model will be created to compare the costs and benefits of three BRCA1/2 mutation testing strategies for patients with HGSEC. Health benefit will be measured in quality adjusted life years (QALYs). Costs in the model will include genetic counselling, genetic tests, breast cancer screening, risk reducing surgeries (RRS), palliative care and cancer treatment for patients and their first and second-degree relatives. QALYs will be calculated per individual and aggregated to provide an incremental cost-effectiveness ratio (ICER).

SECONDARY OUTCOMES:
The proportion of germline and somatic BRCA1 and BRCA2 mutations among patients with HGSEC in Ireland | 78 months
  Descriptive statistics will be calculated to summarize the number of patients with Germline BRCA1/2 mutations, somatic BRCA1/2 mutations and Variants of Unknown Significance (VUS). Counts, ranges and percentages will be used.
Patient and disease characteristics (age, stage, degree of surgical cytoreduction, platinum sensitivity) associated with BRCA1/2 mutated HGSEC compared to BRCA1/2 wild type disease. | 78 months
Differences in treatment patterns between BRCA1/2 mutated and BRCA1/2 wild type HGSEC by examining number of systemic therapies used. | 78 months
Differences in treatment patterns between BRCA1/2 mutated and BRCA1/2 wild type HGSEC by examining use of PARP inhibitor therapy. | 78 months
Differences in treatment patterns between BRCA1/2 mutated and BRCA1/2 wild type HGSEC by examining enrolment in clinical trials | 78 months
Identification of clinical outcomes (response platinum free interval (PFI)) associated with BRCA1/2-mutated HGSEC, as compared to BRCA1/2 wild type disease. | 78 months
Identification of clinical outcomes (progression free survival (PFS)) associated with BRCA1/2-mutated HGSEC, as compared to BRCA1/2 wild type disease. | 78 months
Identification of clinical outcomes (overall survival (OS)) associated with BRCA1/2-mutated HGSEC, as compared to BRCA1/2 wild type disease. | 78 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Bryan Hennessy, Principal Investigator — Beaumont Hospital, Ireland
Locations (5):
- Ireland (5):
  - Mater Misericordiae University Hospital / Mater Private Hospital, Dublin, Leinster
  - St James's Hospital, Dublin, Leinster
  - Bon Secours, Cork, Munster
  - Cork University Hospital, Cork, Munster
  - University Hospital Limerick, Limerick, Munster